CLINICAL TRIAL: NCT01917877
Title: Phase II Study of Bevasizumab in the Management of Acute Radiation-induced and Chemotherapy-induced Pulmonary Fibrosis
Brief Title: Efficiency Study for Acute Radiation-induced and Chemotherapy-induced Pulmonary Fibrosis With Bevasizumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QCH-20030801
Record Dates: First submitted 2013-08-01; First posted 2013-08-07 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-02

CONDITIONS: Pulmonary Fibrosis
Keywords: Becacizumab; pulmonary fibrosis; irradiation; chemotherapy
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Bevacizumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (Experimental): Bevacizumab 7mg/kg iv on day1 and 21, followed by Dexamethasone 10mg iv d 1-10, then 5mg iv d11-15, 2.5mg iv d16-20
  Interventions: Drug: Bevacizumab
- control (Active Comparator): Dexamethasone 10mg iv d 1-10, then 5mg iv d11-15, 2.5mg iv d16-20
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 7mg/kg iv on day1 and 21, followed by Dexamethasone 10mg iv d 1-10, then 5mg iv d11-15, 2.5mg iv d16-20
  Other Names: Avastin (Genentech/Roche)
  Arms: study group
Drug: Dexamethasone — Dexamethasone 10mg iv d 1-10, then 5mg iv d11-15, 2.5mg iv d16-20
  Arms: control

SUMMARY:
Due to the radiosensitivity of the lung, radiation-induced and chemotherapy-induced pneumonitis and pulmonary fibrosis are frequent happened following cancer therapy. It not only compromise cancer treatment, but also influence patient's life qualities and even death. there are no specific treatment modalities for this treatment-induced complication. Bevasizumab (Avastin), a VEGF inhibitor, can attenuate serum high expression VEGF and pulmonary permeability, maybe effective in the control acute pulmonary fibrosis. Patients will be randomized to receive Bevasizumab (7mg/kg iv) on day one and 21, followed by Dexamethasone （10mg iv d 1-10, then 5mg iv d11-15, 2.5mg iv d16-20) or Dexamethasone alone. The thoracic CT, plasma TNF-a, IL-6, VEGF and C-reactive protein are accessed on before treatment, 24 hours after Bevasizumab, 7 days, 4 and 8 weeks. the target sample size is 30 cases.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosed cancer treatment-induced acute pulmonary fibrosis

Exclusion Criteria:

* chronic pulmonary fibrosis and infection-induced pulmonary fibrosis
* active bleeding
* uncontrolled high blood pressure
* unstable systemic disease
* prior exposure to VEGF inhibitor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pulmonary function | up to 8 weeks

SECONDARY OUTCOMES:
thoracic CT scan | up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: youxin ji, md, Principal Investigator — Qingdao Central Hospital
Locations (1):
- Qingdao Central Hospital, Qingdao, Shandong, China